CLINICAL TRIAL: NCT02389738
Title: Brain Interstitium Temozolomide Concentration Pre and Post Regadenoson Administration
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J14155; IRB00045837 (Other: JHM IRB)
Record Dates: First submitted 2015-03-04; First posted 2015-03-17 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Blood Brain Barrier Defect
MeSH Terms: interventions — regadenoson; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BBB disruption with regadenoson (Experimental): This is an exploratory (pilot) study to assess whether Regadenoson can disrupt the BBB, change the barrier permeability, to enhance the temozolomide delivery to brain.
  Five evaluable patients will be studied in this trial. The sample size justification is not based on statistical rationale but clinical affordability. If the investigators detect ≥ 50% increase in temozolomide brain interstitium concentrations after Regadenoson, then the investigators will consider future studies evaluating additional patients.
  Interventions: Drug: Regadenoson; Drug: Temozolomide; Device: Microdialysis catheter

INTERVENTIONS:
Drug: Regadenoson — Regadenoson administration on post-op day 2 after temozolomide administration. Temozolomide plasma and dialysate concentrations will be obtained over 18 hours post temozolomde administration.
  Other Names: Lexiscan
Drug: Temozolomide — Temozolomide administration on post-op day 1 and 2. Temozolomide plasma and dialysate concentrations will be obtained over 18 hours post temozolomde administration.
  Other Names: Temodar
Device: Microdialysis catheter — Microdialysis catheter placement post surgical resection and removed at the bedside after completion of obtaining all dialysate collections.

SUMMARY:
The blood-brain barrier (BBB) is an intricate barrier composed of a variety of efflux pumps, a luminal negative charge, a basal lamina and three distinct cell types: brain endothelial cells, pericytes, and astrocyte foot processes. Specifically, the BBB integrity and degree of permeability is regulated by the capillary endothelial cells in response to astrocytic signals. The strength of intercellular junctions (ex. tight junctions, adherins) amongst endothelial cells also plays a major role in permeability. Therefore, modulation of all these paracellular properties may decrease BBB integrity and thus improve drug penetration to the tumor bed. Previous studies utilizing the vasoactive peptide, Regadenoson, demonstrated transient increase in BBB permeability, allowing a 70kD dextran molecule to enter the brain of rodents. Thus, the investigators propose to evaluate brain interstitium concentrations of temozolomide pre and post Regadenoson using brain microdialysis. If Regadenoson successfully demonstrates effectiveness in disrupting the BBB, it could be of major importance in improving the outcome of patients with a variety of brain tumors and other neurologic illnesses.

DETAILED DESCRIPTION:
Blood brain barrier:

The blood-brain barrier (BBB) is an intricate barricade composed of three distinct cell types: brain endothelial cells, pericytes, and astrocyte foot processes. While molecules that are small and lipophilic may easily traverse the BBB, large (> 180 Daltons) and/or hydrophilic particles require active transport, or receptor mediation. Specifically, the BBB integrity and degree of permeability is regulated by the capillary endothelial cells in response to astrocytic signals. The strength of intercellular junctions (ex. tight junctions, adherins) amongst endothelial cells also plays a major role in permeability. Therefore, modulation of all these paracellular properties may serve a large part in decreasing BBB integrity and thus improving drug penetration to the tumor bed.

Rationale for Regadenoson:

Adenosine may be a plausible means to transiently disrupt the BBB. Adenosine function is regulated by its four structurally related G-protein coupled receptors: A1, A2A, A2B and A3. Specifically, A1 and A2A have high expression levels within the brain. In 2011, Carman et al demonstrated, with the selective A2A receptor agonist, Regadenoson, increased BBB permeability to 70kD Dextran in both mice and rat brains. The large molecule of Dextran was seen in the brain for up to 180 minutes following a single injection in both mice and rats. Studies performed at Johns Hopkins have also demonstrated a transient disruption of the BBB from Regadenoson in rodents by measuring temozolomide concentrations. The investigators found that brain/plasma concentrations in rats post Regadenoson resulted in a 1.6 fold increase of temozolomide compared to temozolomide given alone in normal rat brains. Future animal studies will evaluate varied chemotherapy agents within the brain and brain tumor with and without Regadenoson.

Currently, Regadenoson is approved by the US Food and Drug Administration as a coronary vasodilator, for myocardial perfusion imaging in patients with suspected myocardial coronary artery disease. Single-photon emission computed tomography (SPECT) imaging performed with 99mTc-sestamibi radiotracer is used to measure coronary blood flow both at rest and stress conditions with Regadenoson. While the adverse event profile is similar to adenosine, the most common side effects of Regadenoson are flushing, chest pain, dyspnea and headaches.

Intracerebral Microdialysis:

Plasma drug concentration measurements are an unreliable method to assess delivery of drugs across the BBB. In contrast, intracerebral microdialysis monitoring allows for approximate measurements within extracellular fluid (ECF) sampling of the brain. Microdialysis placement within the brain is not a novel technique and has been utilized routinely in the intensive care unit setting to measure brain metabolism by sampling of ECF of traumatic brain injury patients. Microdialysis catheters are now FDA approved and are being placed routinely with intracranial pressure monitors. This method allows for continuous measurement of ECF within a tumor or normal tissue. The dialysis probe has a semipermeable membrane which is less than 1 mm in diameter into which two sections of microcatheter are fused. Previous studies have demonstrated the feasibility of keeping the catheters in place of critically injured patients for up to 2 weeks. When placed at the time of surgical resection, the microcatheters are sterotactically implanted, placing the probe within the desired brain and/or tumor region. Externally, the catheter is connected to a syringe pump, which delivers a low flow rate (µl/min) of continuous perfusion fluid (Lactated Ringers or artificial CSF) and dialysate is collected in a microvial from the outlet tube. This sterile, single use catheter is minimally invasive and developed to achieve optimal diffusing characteristics similar to passive diffusion of a capillary blood vessel. Just as in the function of brain capillary vessel, water, inorganic ions and small organic molecules freely diffuse across the membrane of the probe, whereas proteins and protein bound compounds are impermeable. Additionally, lipophilic compounds are poorly recovered.

Use of Intracerebral Microdialysis to Quantitate temozolomide Concentrations Temozolomide is a FDA approved oral alkylating agent used in upfront and relapsed therapy of adult and pediatric patients with high grade glioma. While temozolomide (TMZ) with radiotherapy has assisted with improving overall survival rates of high grade gliomas, previous studies have proven approximately only 20% of the drug crosses the BBB after peripheral administration. The peak concentration of TMZ in the brain has been shown to be approximately 1-2 hours after ingestion. Once ingested, TMZ undergoes degradation from its prodrug form to the highly reactive alkylating agent, methyl-triazenyl imidazole carboxamide (MTIC). Previous studies have utilized brain microdialysis catheters to measure TMZ brain interstitium levels post primary or metastatic brain resection/biopsy. Both serum and dialysates were collected at 30 minute time intervals and analyzed to quantitate TMZ drug delivery to the tumor bed and surrounding tissue yet due to drug stability issues, MTIC concentrations were not feasible for measurement in the microdialysis setting. Thus, the investigators propose to measure TMZ concentrations pre and post Regadenoson administration with the hypothesis that transient BBB disruption will result in improved drug efficacy to the brain interstitium and tumor bed. If gross total resection cannot be achieved two microdialysis catheters will be placed after resection. One microdialysis catheter will be placed in the MRI enhancing tumor area and one catheter will be placed in a non-enhancing area, allowing for later assessment of the degree of BBB permeability both in the tumor and normal brain. These studies will be beneficial to evaluate the role of increasing temozolomide delivery in an effort to further increase tumor cytotoxicity and progression-free survival in such an aggressive tumor.

Use of Intracerebral Microdialysis to Quantitate Markers of Neuroinflammation Previous studies have demonstrated that patients with increased inflammatory cytokines from medical illnesses exhibit increased rates of depression. Both chronic and acutely elevated levels of inflammatory cytokines can result in the development of neuropsychiatric dysfunction, including cognitive slowing, inattention, or depression. Specifically, Dowlati et al concluded from a meta-analytic study that a small proportion of patients with idiopathic major depressive disorder exhibited increased serum cytokine levels. Thus, the investigators propose to quantitate markers of neuroinflammation and oxidative stress in collected dialysate, with the hypothesis that variance in these levels may correlate with affective and/or cognitive dysfunction.

Risks of Microdialysis:

These studies will be a novel investigation in the use of brain microdialysis to measure TMZ concentration in the post-operative setting with combinational administration of Regadenoson and temozolomide. To minimize risks post-surgical resection or biopsy, patients will only receive temozolomide 150mg/m2 twice, which is less than half the standard 5 day course administered during maintenance therapy for malignant glioma post radiation therapy. In addition, therapy will be given for only two days in the ICU setting, with minimal tumor toxicity anticipated with a suboptimal treatment dose over a short duration.[ The procedures involved with the insertion and removal of the dialysis probe can be performed with minimal injury at the time of surgery.[18,19] Although insertion of the microdialysis probe could conceivably disrupt the BBB, this has not proven to be problematic, as demonstrated by rapid normalization of the BBB after placement, allowing for equilibration and minimization of artifact.[20-22] Although it can be safely performed, microdialysis is nevertheless an invasive surgical procedure with a small risk of bleeding at the site of insertion and discomfort for the patient. The previous study which evaluated brain interstitium concentrations of TMZ evaluated dialysate samples from seven patients. All of the patients tolerated placement of the catheters and collection of the dialysate samples well, yet 1 patient developed several grade 3 and 4 neurologic adverse events whose etiologies remain unclear. All of the neurologic deficits improved without completely resolving.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Diagnosis of recurrent high grade glioma confirmed by frozen pathology intra-operatively
* Patients with planned surgical debulking or biopsy
* Karnofsky performance status (KPS) ≥ 60%
* Mini Mental Status Exam ≥ 15
* Adequate hepatic function
* Total bilirubin ≤ 1.8 mg/dL
* Serum levels of aspartate aminotransferase ≤ 3x the institutional upper limit of normal
* Adequate renal function
* Serum creatinine ≤ 1.5mg/dL
* Adequate bone marrow function
* ANC ≥ 1500 cells/mm3
* Platelet count ≥ 100,000 cells/mm3

Exclusion Criteria:

* Currently receiving chemotherapy, or radiation therapy
* Allergic to temozolomide
* Pregnant or breast-feeding
* Have a serious medical or psychiatric illness or social situation that could interfere with catheter placement or monitoring
* Prior use of VEGF or VEGFR-targeted therapy
* Use of medications: Vincristine, Vinblastine, Rifampin, Opioid's, Antidepressants within the past 24 hours
* Use of investigational agents within the past 4 weeks
* NCI CTC Grade 3 or greater baseline neurologic symptoms
* History of cardiac disease:
* Atrial fibrillation or uncontrolled tachyarrhythmia, or advanced atrioventricular block (second or third degree heart block)
* History of sinus node dysfunction
* History of symptomatic sinus bradycardia or recorded (heart rate <40/minute)
* Use of dipyridamole, dipyridamole-containing medications
* Any history of coronary heart disease defined by prior myocardial infarction or ischemia on cardiac stress testing or coronary stenosis ≥50% severity
* Moderate or severe aortic stenosis
* Uncontrolled hypertension (BP >200/110)
* Decompensated or inadequately controlled congestive heart failure.
* Acute pulmonary embolism
* Acute myocarditis or pericarditis
* Acute aortic dissection
* Severe pulmonary hypertension
* Hypertrophic obstructive cardiomyopathy
* Electrolyte abnormalities
* Unexplained chest pain that may be anginal in nature
* Use of sublingual nitroglycerin
* History of Regadenoson hypersensitivity
* Known symptomatic hypotension, uncontrolled hypertension within 30 days
* History of moderate to severe bronchospastic lung disease (including moderate to severe asthma)
* Use of aminophylline in the last 24 hours
* Use methylxanthine or caffeine in the last 12 hours
* Contraindication to adenosine (e.g., bronchoconstrictive/bronchospastic disease)
* Use of potassium supplements or potassium sparing medications in the past 24 hours
* Any patient not deemed medically stable by a physician
* Recent history of illicit drug use (past 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2018-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Grossman, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- BBB Disruption With Regadenoson: This is an exploratory (pilot) study to assess whether Regadenoson can disrupt the BBB, change the barrier permeability, to enhance the temozolomide delivery to brain.
  Five evaluable patients will be studied in this trial. The sample size justification is not based on statistical rationale but clinical affordability. If the investigators detect ≥ 50% increase in temozolomide brain interstitium concentrations after Regadenoson, then the investigators will consider future studies evaluating additional patients.
  Regadenoson: Regadenoson administration on post-op day 2 after temozolomide administration. Temozolomide plasma and dialysate concentrations will be obtained over 18 hours post temozolomde administration.
  Temozolomide: Temozolomide administration on post-op day 1 and 2. Microdialysis catheter: Microdialysis catheter placement post surgical resection Temozolomide plasma and dialysate concentrations will be obtained over 18 hours post temozolomde administration.
Period: Overall Study
Arm/Group | BBB Disruption With Regadenoson
Started | 6
Completed | 5
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- BBB Disruption With Regadenoson: This is an exploratory (pilot) study to assess whether Regadenoson can disrupt the BBB, change the barrier permeability, to enhance the temozolomide delivery to brain.
  Five evaluable patients will be studied in this trial. If the investigators detect ≥ 50% increase in temozolomide brain interstitium concentrations after Regadenoson, then the investigators will consider future studies evaluating additional patients.
  Regadenoson: Regadenoson administration on post-op day 2 after temozolomide administration. Temozolomide plasma and dialysate concentrations will be obtained over 18 hours post temozolomde administration.
  Temozolomide: Temozolomide administration on post-op day 1 and 2. Temozolomide plasma and dialysate concentrations will be obtained over 18 hours post temozolomde administration.
  Microdialysis catheter: Microdialysis catheter placement post surgical resection and removed at the bedside after completion of obtaining all dialysate collections.
Arm/Group | BBB Disruption With Regadenoson
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 51 [32 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in AUC0-18 of the Temozolomide Concentration (AUC-T) in Brain Interstitium Before and After Regadenoson Infusion
Description: The AUC-T for each day will be estimated by the trapezoid rule, based on the number of time points available for the particular evaluable patient. The PK variables will be tabulated and descriptive statistics calculated pre and post Regadenoson. The difference of AUCs will be summarized by mean and standard deviation or median and range if there is large variation from patient to patient. Means and standard deviation or mean and range will be presented for Cmax and AUC(inf) for each group. Graphic method will be used to display the difference for individual patient and all five patients.
Time Frame: 18 hours post temozolomide administration
Measure: Mean (Full Range); unit: percentage of AUC
Groups:
- BBB Disruption With Regadenoson: This is an exploratory (pilot) study to assess whether Regadenoson can disrupt the BBB, change the barrier permeability, to enhance the temozolomide delivery to brain.
  Five evaluable patients will be studied in this trial. The sample size justification is not based on statistical rationale but clinical affordability. If the investigators detect ≥ 50% increase in temozolomide brain interstitium concentrations after Regadenoson, then the investigators will consider future studies evaluating additional patients.
  Regadenoson: Regadenoson administration on post-op day 2 after temozolomide administration. Temozolomide plasma and dialysate concentrations will be obtained over 18 hours post temozolomde administration.
  Temozolomide: Temozolomide administration on post-op day 1 and 2. Microdialysis catheter: Microdialysis catheter placement post surgical resection. Temozolomide plasma and dialysate concentrations will be obtained over 18 hours post temozolomde administration.
Arm/Group | BBB Disruption With Regadenoson
Number analyzed (Participants) | 5
percentage of AUC
  Temozolomide alone AUC brain/plasma | 19.1 [3.3 to 31.5]
  Temozolomide/Regadenoson AUC brain/plasma | 18.0 [7.5 to 27.5]

2. Secondary Outcome: Evaluation of Relationaship Between Cognitive/Mood Disorders and Expression of Biochemical Markers Post-op Day 1
Description: The study of collecting biochemical markers of glioma with correlation to current or past cognitive/mood disorders with Montgomery-Asberg. Biomarkers will be obtained post-op day 1 from dialysate collections and later identified and quantified.
Time Frame: 24 hours post-op
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- BBB Disruption With Regadenoson: This is an exploratory (pilot) study to assess whether Regadenoson can disrupt the BBB, change the barrier permeability, to enhance the temozolomide delivery to brain.
  Five evaluable patients will be studied in this trial. The sample size justification is not based on statistical rationale but clinical affordability. If the investigators detect ≥ 50% increase in temozolomide brain interstitium concentrations after Regadenoson, then the investigators will consider future studies evaluating additional patients.
  Regadenoson: Regadenoson administration on post-op day 2 after temozolomide administration.
  Temozolomide: Temozolomide administration on post-op day 1 and 2.
  Microdialysis catheter: Microdialysis catheter placement post surgical resection and removed at the bedside after completion of obtaining all dialysate collections obtained over 18 hours post temozolomde administration.
Arm/Group | BBB Disruption With Regadenoson
All-Cause Mortality (participants affected / at risk) | 5/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes